CLINICAL TRIAL: NCT02731638
Title: Mycotic Antimicrobial Localized Injection for Treatment of Corneal Ulcers
Acronym: MALIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-17989
Record Dates: First submitted 2016-03-14; First posted 2016-04-07 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Corneal Ulcer; Fungal Keratitis
Keywords: cornea; ulcer; fungal; keratitis
MeSH Terms: conditions — Corneal Ulcer; Corneal Diseases; Ulcer; Keratitis | interventions — Natamycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrastromal voriconazole plus natamycin (Experimental): Intrastromal voriconazole plus standard of care topical treatment for fungal keratitis
  Interventions: Drug: Intrastromal voriconazole; Drug: Natamycin
- Natamycin alone (Active Comparator): Standard of care topical treatment for fungal keratitis
  Interventions: Drug: Natamycin

INTERVENTIONS:
Drug: Intrastromal voriconazole — Subjects will receive three intrastromal voriconazole injections over 10 days. Intrastromal voriconazole injection is a routine procedure performed by Aravind Eye Hospital for fungal keratitis.
  Arms: Intrastromal voriconazole plus natamycin
Drug: Natamycin — Subjects will receive topical 5% natamycin drops hourly for 3 days.

SUMMARY:
Mycotic Antimicrobial Localized Injection (MALIN) is a randomized, masked, two-arm clinical trial investigating intrastromal voriconazole in the treatment of fungal corneal ulcers. There is currently little evidence to guide the treatment of fungal keratitis beyond topical anti-fungal drops, though intrastromal voriconazole and oral antifungal treatments are used as well. This study will provide evidence to guide the treatment of fungal keratitis in the future. The purpose of this study is to determine differences in microbiological cure for 3-day repeat cultures between different antifungal treatments. For this study, there will be 1:1 randomization to one of these two treatment groups: 1) topical natamycin plus intrastromal voriconazole injection or 2) topical natamycin alone.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial to determine whether intrastromal voriconazole improves outcomes in fungal keratitis. Patients presenting to the Aravind Eye Hospitals in Pondicherry, India for treatment of fungal keratitis will be recruited for the proposed study. Approximately 70 patients will be enrolled in the study. Subjects presenting with fungal keratitis will be randomized to receive topical natamycin plus intrastromal voriconazole or to receive topical natamycin alone. Subjects may also receive oral antifungals after day 3 at the discretion of the treating clinician. All study subjects will be followed for 3 months to evaluate response to treatment.

Investigators from the University of California, San Francisco (UCSF) will assist Aravind Eye Hospital with the study design, implementation, and analysis of the research, and will help fund the study. The investigators will visit Aravind to help with the study implementation. UCSF will play an important role in this study by assisting with the study design, implementation, analysis, and funding.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe corneal ulcer that is smear positive for filamentous fungus
* Pinhole visual acuity worse than 20/70 in affected eye
* Basic understanding of the study as determined by the physician
* Commitment to return for follow up visits

Exclusion Criteria:

* Gram stain positive for bacteria or evidence of other concomitant infection (i.e. herpes, acanthamoeba)
* Impending or frank perforation at recruitment
* Involvement of sclera at presentation
* Non-infectious or autoimmune keratitis
* History of corneal transplantation or recent intraocular surgery
* No light perception in the affected eye
* Pinhole visual acuity worse than 20/200 in the unaffected eye
* Pregnant women
* Participants who are decisionally and/or cognitively impaired

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rose-Nussbaumer, MD, Principal Investigator — Stanford University
Locations (2):
- Francis I. Proctor Foundation at UCSF, San Francisco, California, United States
- Aravind Eye Hospitals, Pondicherry, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be input into a database using double data entry at UCSF. Data will be stored at UCSF for about 10 years.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrastromal Voriconazole Plus Natamycin | Natamycin Alone
Started | 35 | 35
Completed | 29 | 26
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrastromal Voriconazole Plus Natamycin | Natamycin Alone | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [42 to 60] | 55 [41 to 62] | 55 [43 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 26 | 18 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 35 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 35 | 35 | 70
Occupation [Count of Participants; unit: Participants]
  Agriculture | 11 | 15 | 26
  Non-Agriculture | 22 | 17 | 39
  Unknown | 2 | 3 | 5
Trauma [Count of Participants; unit: Participants]
  Stick | 7 | 3 | 10
  Leaf | 2 | 1 | 3
  Finger | 0 | 1 | 1
  Dust | 3 | 4 | 7
  Mud | 4 | 4 | 8
  Insect | 5 | 1 | 6
  Other | 4 | 9 | 13
  Unknown object | 0 | 2 | 2
  No trauma | 10 | 10 | 20
Affected Eye [Count of Participants; unit: Participants]
  Right | 15 | 17 | 32
  Left | 20 | 18 | 38
Visual Acuity, logMAR [Median (Inter-Quartile Range); unit: logMAR] — Visual acuity in logarithm of the minimum angle of resolution (logMAR) units
  logMAR | 1.7 [1.6 to 1.8] | 1.7 [1.6 to 1.8] | 1.7 [1.6 to 1.8]
Ulcer location [Count of Participants; unit: Participants]
  Central | 30 | 32 | 62
  Peripheral | 5 | 3 | 8
Hypopyon size (mm) [Count of Participants; unit: Participants]
  None | 16 | 13 | 29
  <0.5mm | 6 | 7 | 13
  ≥0.5mm | 13 | 15 | 28
Ulcer depth, measured in % depth [Count of Participants; unit: Participants]
  >0-33% | 13 | 10 | 23
  >33-67% | 11 | 16 | 27
  >67-100% | 11 | 9 | 20
Culture Results [Count of Participants; unit: Participants]
  Fusarium species | 8 | 11 | 19
  Aspergillus species | 7 | 10 | 17
  Curvularia species | 4 | 0 | 4
  Exserohilum species | 1 | 1 | 2
  Unidentified hyaline | 3 | 2 | 5
  Unidentified dematiaceous | 3 | 5 | 8
  Fungal culture negative | 8 | 5 | 13
  Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Culture Positivity at Day 3 Using Potassium Hydroxide (KOH) Wet Mount to Test for Fungus
Description: Number of of participants with positive fungal cultures at 3 days
Time Frame: 3 days
Population: 3-day culture results missing for one participant in the Natamycin group
Measure: Count of Participants; unit: Participants
Arm/Group | Intrastromal Voriconazole Plus Natamycin | Natamycin Alone
Number analyzed (Participants) | 35 | 34
Participants | 14 | 11
Statistical Analysis 1: Comparison: Intrastromal Voriconazole Plus Natamycin vs Natamycin Alone; Test type: Superiority; p = 0.26, Regression, Logistic; Bias-corrected logistic regression, accounting for baseline culture status; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.65 to 5.23]

2. Secondary Outcome: Best Spectacle-corrected Visual Acuity, as Measured by a Refractionist
Description: Best spectacle-corrected visual acuity using calibrated Original Series Early Treatment Diabetic Retinopathy Study eye charts and recorded as number of letter read.
Time Frame: 3 weeks and 3 months
Population: 3-week visual acuity data was available for 65 people: 33 in the ISV group (2 lost to follow-up) and 32 in the Natamycin only group (3 lost of follow-up). 3-month visual acuity data was available for 58 people: 30 in the ISV group (5 lost to follow-up) and 28 in the Natamycin only group (7 lost to follow-up).
Measure: Mean (Standard Deviation); unit: logarithm of the minimum angle (logMAR)
Arm/Group | Intrastromal Voriconazole Plus Natamycin | Natamycin Alone
Number analyzed (Participants) | 33 | 32
logarithm of the minimum angle (logMAR)
  3 weeks | 1.39 (0.59) | 1.23 (0.65)
  3 months: number analyzed (Participants) | 30 | 28
  3 months | 1.30 (0.60) | 1.28 (0.66)
Statistical Analysis 1: Comparison: Intrastromal Voriconazole Plus Natamycin vs Natamycin Alone; Test type: Superiority; p = 0.25, Regression, Linear; Coefficient = 1.6, 95% CI 2-sided [-1.2 to 4.4] — Positive coefficients of the logMAR value indicated worsened visual acuity
Statistical Analysis 2: Comparison: Intrastromal Voriconazole Plus Natamycin vs Natamycin Alone; Test type: Superiority; p = 0.75, Regression, Linear; Coefficient = 0.5, 95% CI 2-sided [-2.6 to 3.6] — Positive coefficients of the logMAR value indicate worsened visual acuity

3. Secondary Outcome: Scar Size
Description: Scar size, geometric mean
Time Frame: 3 weeks and 3 months
Population: 3-week scar size data was available for 42 people: 24 in the ISV group (2 lost to follow-up [LTF], 9 unable to assess) and 18 in the Natamycin only group (3 LTF, 14 unable to assess). 3-month scar size data was available for 29 people: 16 in the ISV group (5 LTF, 14 unable to assess) and 13 in the Natamycin only group (7 LTF, 15 unable to assess).
Measure: Mean (Standard Deviation); unit: millimeters squared
Arm/Group | Intrastromal Voriconazole Plus Natamycin | Natamycin Alone
Number analyzed (Participants) | 24 | 18
millimeters squared
  3 Weeks | 4.8 (1.2) | 4.1 (1.3)
  3 Months: number analyzed (Participants) | 16 | 13
  3 Months | 4.9 (1.2) | 4.5 (1.1)

4. Secondary Outcome: Number of Participants With Scar Depth at the Anterior Third, Middle Third, and Posterior Third of the Cornea
Description: Number of participants with scar depth at the anterior third (0-33% depth), middle third (>33-67% depth), and posterior third (>67-100% depth) of the cornea, as measured on slit lamp exam.
Time Frame: 3 weeks and 3 months
Population: 3-week scar depth data was available for 40 people: 24 in the ISV group (2 lost to follow-up [LTF], 9 unable to assess) and 16 in the Natamycin only group (3 LTF, 16 unable to assess). 3-month scar depth was available for 29 people: 16 in the ISV group (5 LTF, 14 unable to assess) and 13 in the Natamycin only group (7 LTF, 15 unable to assess).
Measure: Count of Participants; unit: Participants
Arm/Group | Intrastromal Voriconazole Plus Natamycin | Natamycin Alone
Number analyzed (Participants) | 24 | 16
Participants
  3 Weeks: Anterior third | 9 | 13
  3 Weeks: Middle third | 8 | 2
  3 Weeks: Posterior third | 7 | 1
  3 Months: number analyzed (Participants) | 16 | 13
  3 Months: Anterior third | 6 | 7
  3 Months: Middle third | 5 | 2
  3 Months: Posterior third | 5 | 4

5. Other Pre Specified Outcome: Corneal Neovascularization
Description: As measured by clinical examination and slit lamp photographs.
Time Frame: 3 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Quality of Life, Measured by the Indian Vision Function Questionnaire (IND-VFQ)
Time Frame: 3 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Corneal Thinning, as Measured by Pachymetry and OCT
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Corneal Topography, as Measured by a Non-contact Imaging Topographer
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intrastromal Voriconazole Plus Natamycin | Natamycin Alone
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 16/35 | 15/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intrastromal Voriconazole Plus Natamycin (N=35) | Natamycin Alone (N=35)
Endophthalmitis (Eye disorders) | 0 | 2
Glaucoma (Eye disorders) | 4 | 2
Hypopyon (Eye disorders) | 3 | 0
Medication Reaction (Eye disorders) | 0 | 1
Nonhealing Ulcer (Eye disorders) | 3 | 0
Perforation (Eye disorders) | 8 | 3
Progressive Corneal Thinning (Eye disorders) | 1 | 0
Therapeutic Penetrating Keratoplasty (Eye disorders) | 14 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT02731638/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT02731638/SAP_001.pdf